CLINICAL TRIAL: NCT02906748
Title: Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology
Brief Title: Parathyroid Auto-transplantation: Prospective Randomized Trial of the Personalized Site
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Gaosong Wu, Doctor, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PA in Tongji Hospital
Record Dates: First submitted 2016-09-12; First posted 2016-09-20 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Parathyroid Autologous Transplantation
Keywords: parathyroid autografting; thyroidectomy; survival rate; hypoparathyroidism
MeSH Terms: conditions — Hypoparathyroidism | interventions — Injections

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- new site for parathyroid auto-graft (Experimental): choose the site fairly close to the antecubital vein for parathyroid auto-transplantation
  Interventions: Procedure: injection with a syringe in new-site for parathyroid autografting
- traditional parathyroid autograft (Active Comparator): choose not intensely close to antecubital vein for parathyroid auto-transplantation
  Interventions: Procedure: injection with a syringe in traditional site for parathyroid autografting

INTERVENTIONS:
Procedure: injection with a syringe in new-site for parathyroid autografting — new-site for parathyroid autografting, close to the antecubital vein
  Other Names: parathyroid autotransplantation; parathyroid auto-implantation; parathyroid auto-graft
  Arms: new site for parathyroid auto-graft
Procedure: injection with a syringe in traditional site for parathyroid autografting — traditional-site for parathyroid autografting,not intensively close to the antecubital vein
  Arms: traditional parathyroid autograft

SUMMARY:
The functional parathyroid auto-transplantation (PA) could release parathyroid hormone (PTH) into the circulatory system of the body through the capillaries. But when parathyroid glands were auto-grafted in the sternocleidomastoid muscle, it would be inconvenient to detect PTH to examine whether the graft functions. So the investigators took the forearm as the aim place for auto-transplantation, either subcutaneous or brachioradialis, with its relatively fixed - antecubital vein blood test which is simple. The survival criteria is assumed as the PTH gradient of 1.5 times or greater through comparing the bilateral PTH value in grafted and not-grafted forearm.

ELIGIBILITY:
Inclusion Criteria:

* patients with indications for PA treatment during cervical surgery

Exclusion Criteria:

* patients suffering secondary hypoparathyroidism with forearm fistulization

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
parahthyroid hormone gradient by comparing between grafted and non-grafted forearm | 1 months, 3 months and 6 months
  The survival criteria is that the gradient of parathyroid hormone reaches 1.5 time or greater by comparing between grafted and non-grafted forearm

SECONDARY OUTCOMES:
hypoparathyroidism: parathyroid hormone less than 15pg/ml(range from 15 to 65pg/ml) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gaosong Wu, PhD, Study Director — Department of Thyroid and Breast Surgery Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

REFERENCES:
- [Derived] Cui Q, Kong D, Li Z, Wang K, Zhang D, Tang J, Liao X, Yuan Q, Gong Y, Wu G. Parathyroid autotransplantation at a novel site for better evaluation of the grafted gland function: study protocol for a prospective, randomized controlled trial. Trials. 2019 Jan 31;20(1):96. doi: 10.1186/s13063-019-3195-9. PMID 30704522